CLINICAL TRIAL: NCT06355336
Title: Patient Reported Data on Prostate Cancer Diagnosis, Management, and Outcome: Real World Prostate Cancer Registry
Brief Title: Real World Prostate Cancer Registry
Acronym: RWPCR
Status: Recruiting | Type: Observational
Sponsor: Cincinnati Cancer Advisors (Network)
Responsible Party: Sponsor
Other Study IDs: CCA/IRN-24-001
Record Dates: First submitted 2024-03-21; First posted 2024-04-09 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Prostate cancer is the most common cancer diagnosed in men in the USA with 268,490 cases diagnosed in 2022 constituting 27% of male cancers and 34,500 deaths (11%) occurred in same year.1 Prostate cancer is a very heterogeneous disease that has different presentations, molecular and pathological features, stages, and disease biology. The treatment options are dependent on the disease stage, its features, and the patient's condition and preferences. The disease outcome also varies significantly due to the previous heterogeneity of the features in addition to other social determinants of health.

Therefore, it is critical to obtain real-world data that reflects the actual patterns of prostate cancer presentation, work up, management, and outcome. Real World Prostate Cancer Registry (RWPCR) aims at compiling real world data from patients presented with prostate cancer in the tristate area. The data collection will be prospective and longitudinal including patients' demographics and disease characteristics, work up, management, and outcome.

DETAILED DESCRIPTION:
Real World Prostate Cancer Registry (RWPCR) aims at compiling real world data from patients presented with prostate cancer in the tristate area. The data collection will be prospective and longitudinal including patients' demographics and disease characteristics, work up, management, and outcome.

Primary Objectives: Describing the patterns of prostate cancer presentation, management, and outcome in the studied population Identify any impact of the compiled variables on treatment selection, work up and outcome.

Secondary Objectives: Identify any gaps and variations in the delivery of care, challenges and needs to optimize management of the disease and improve patient's outcome.

Improve awareness and facilitate enrollment into clinical trials and research studies.

Data will be collected directly from patients. This data will be collected over 10 years with three years of enrollment and seven years of follow-up. Patients provide e-consent and then get login credentials to complete the e-forms which can be edited and updated by the patient. 6 monthly reminders will be sent to the patients to complete 6 monthly follow-ups

Research staff may contact patients to offer opportunities to participate in clinical trials if eligible. A gift card will be provided to the patient for the initial survey submission. A gift card will also be provided to the patient for each 6 month follow up submission.

ELIGIBILITY:
Inclusion Criteria:

All patients with pathologically confirmed primary prostate cancer

Diagnosis since January 1st, 2023

Acceptance to sign the consent form

18 years old or older

Resident of Ohio, Kentucky or Indiana

Exclusion Criteria:

Having diagnosis of other cancer except squamous cell cancer of the skin

Refusal to sign a consent form.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Residents of Ohio, Kentucky or Indiana
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-03-18 (Actual); Primary Completion 2034-03-18 (Estimated); Study Completion 2034-03-18 (Estimated)

PRIMARY OUTCOMES:
To determine practice patterns for prostate cancer in the region. | 10 years
  Descriptive analysis of the disease risk groups, disease stages, and type of treatments provided to the patients (radiation, surgery, hormonal therapy).

SECONDARY OUTCOMES:
To determine progression free survival and overall survival of patients. | 10 years
  Percentage of patients participating in clinical trials.
Prevalence of long term complications of prostate cancer treatment. | 10 years
  Specifically urine incontinence and erectile dysfunction.

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Cancer Advisors, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel RL, Miller KD, Fuchs HE, Jemal A. Cancer statistics, 2022. CA Cancer J Clin. 2022 Jan;72(1):7-33. doi: 10.3322/caac.21708. Epub 2022 Jan 12. PMID 35020204